CLINICAL TRIAL: NCT03223311
Title: "Percutaneous Axillary Access in the Endovascular Treatment of Thoracoabdominal Aortic Pathology"
Brief Title: "Percutaneous Axillary Access in the Endovascular Treatment of Thoracoabdominal Aortic Pathology" (PAXA)
Acronym: PAXA
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Bertoglio Luca, Principal Investigator, IRCCS San Raffaele
Other Study IDs: PAXA/31/OSR
Record Dates: First submitted 2017-07-07; First posted 2017-07-21 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Thoracoabdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Since the development of custom-made fenestrated and branched endografts a novel therapeutic option for the management of thoracoabdominal and para-renal aortic aneurysms was made accessible. Because of the design of these branched endografts, an arterial vascular access from the upper limb is required to allow selective catheterization of the branch component and the respective target vessel (celiac trunk, superior mesenteric artery, renal artery).2

DETAILED DESCRIPTION:
Primary end-point is to evaluate the requirement of upper extremity arterial access (UEA) retrospectively in the cohort of patients with thoracoabdominal aortic aneurysms treated by means fenestrated and/or branched endografts in Vascular surgery San Raffaele Hospital between 2013 and 2017, and prospectively in the next 50 patients that will be treated between 2017 and 2020.

Secondary end-point is an anatomical evaluation of the different sites available for UEA(upper extremity arterial access ) based on pre-operative imaging studies.

Materials and methods:

The investigators review a prospectively compiled Microsoft Office Excel database with the procedural details of the 34 patients treated at Vascular surgery of San Raffaele Hospital between October 2013 and March 2017 by means of total endovascular thoracoabdominal aortic aneurysm repair and of those of the next 50 patients who will be treated until December 2020. All patients in which an UAE (upper extremity arterial access ) is employed will be identified together with the side (left/right) and site (proximal/distal axillary artery, brachial artery) of vascular access. Furthermore, the pre-operative contrast-enhanced computed tomography scans (CTA) of all patients, stored in the hospital PACS, will be analyzed on the dedicated workstation with OsiriX software (Pixmeo sarl, Bernex, Switzerland) currently employed at Vascular surgery of San Raffaele Hospital for imaging assessment.

Requirement of an UEA(upper extremity arterial access ) during the procedure is extrapolated from the corresponding field of the available database and reported together with side and site of access and reason for the employment of UEA (upper extremity arterial access ) and for its location.

Multi-planar, curved and 3D reconstructions of each patient CTA will be analyzed and the following measurements recorded:

1. patency of both potential upper extremity access vessels (right/left subclavian artery);
2. diameter of the proximal axillary artery on both sides;
3. diameter of the distal axillary artery on both sides;
4. presence of calcifications on the proximal axillary artery on both sides;
5. presence of calcifications on the distal axillary artery on both sides;
6. arterial tortuosity index on both sides: measured as the ratio between the axillary artery length measured on curved reconstruction and its length measured on 3D reconstruction.

All the assessed variables will be prospectively recorded in a Microsoft Office Excel database together with patients' weight, height, age and gender.

All patients involved in the retrospective part of the study have already signed informed consent for data collection and analysis at hospital admission.

The 50 patients that will be enrolled until December 2020 will also sign an "ad hoc" consents, specific for this study.

Sensitive patient information will not be available during data analysis. The clinical study will be carried out according to the ethical principles of the Declaration of Helsinki and following the active regulations on observational studies.

Analysis:

Patients characteristics and anatomical data on UEAs(upper extremity arterial access) will be analyzed on Wizard Statistics software to investigate the presence of statistically significant Pearson correlations among the identified variables.

The extracted data and their relevant clinical and procedural implications will be submitted for publication in peer-reviewed scientific journals focused on the field of vascular and endovascular surgery.

ELIGIBILITY:
Inclusion criteria:

• Patient undergoing total endovascular treatment of thoracoabdominal pathology at San Raffaele Hospital in between October 2013 and December 2020.

Exclusion criteria:

• Incomplete imaging quality not including the arterial segments to be studied (axillary and brachial artery).

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patient undergoing total endovascular treatment of thoracoabdominal pathology
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Use of upper extremity access in endovascular repair of thoracoabdominal aortic aneurysms | between 2013 and 2020
  * Endovascular graft design : branched / fenestrated
  * Employment of UEA(upper extremity arterial access ) during TAAA endovascular repair: yes / no
  * Side of UEA(upper extremity arterial access ) cannulation (left / right)
  * Site of UEA(upper extremity arterial access ) cannulation:proximal axillary artery / distal axillary artery / upper brachial artery.
  * Size of percutaneuos access sheath employed measured in French - Fr
  * Number of percutaneuos access vessel closure devices employed
  * Access closure specific outcome: primary success / secondary success / failure As reported on patients' charts and operative report

SECONDARY OUTCOMES:
Upper extremity access vascular anatomy | between 2013 and 2017.
  * UEA(upper extremity arterial access ) vessel patency: yes / no
  * Diameter of proximal axillary artery measured in Millimeters ( mm)
  * Diameter of distal axillary artery measured in Millimeters (mm)
  * Presence of calcifications at UEA(upper extremity arterial access ): none / < 50% / > 50%.
  * Tortuosity index reported as bare number, defined as the ratio between the axillary artery length measured on curved centerline reconstruction and its length measured on 3D reconstruction.
  As measured at preoperative contrast-enhanced CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Luca Bertoglio, MD, Principal Investigator — SAn Raffaele Hospital
Locations (1):
- San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alvarez-Tostado JA, Moise MA, Bena JF, Pavkov ML, Greenberg RK, Clair DG, Kashyap VS. The brachial artery: a critical access for endovascular procedures. J Vasc Surg. 2009 Feb;49(2):378-85; discussion 385. doi: 10.1016/j.jvs.2008.09.017. Epub 2008 Nov 22. PMID 19028057
- [Result] Chuter TA, Rapp JH, Hiramoto JS, Schneider DB, Howell B, Reilly LM. Endovascular treatment of thoracoabdominal aortic aneurysms. J Vasc Surg. 2008 Jan;47(1):6-16. doi: 10.1016/j.jvs.2007.08.032. Epub 2007 Nov 5. PMID 17980540
- [Derived] Bertoglio L, Grandi A, Melloni A, Kahlberg A, Melissano G, Chiesa R. Percutaneous AXillary Artery (PAXA) Access at the First Segment During Fenestrated and Branched Endovascular Aortic Procedures. Eur J Vasc Endovasc Surg. 2020 Jun;59(6):929-938. doi: 10.1016/j.ejvs.2020.01.027. Epub 2020 Feb 20. PMID 32089506
- [Derived] Bertoglio L, Mascia D, Cambiaghi T, Kahlberg A, Melissano G, Chiesa R. Percutaneous axillary artery access for fenestrated and branched thoracoabdominal endovascular repair. J Vasc Surg. 2018 Jul;68(1):12-23. doi: 10.1016/j.jvs.2017.09.053. Epub 2018 Mar 1. PMID 29503006